CLINICAL TRIAL: NCT04995536
Title: A Phase I Study of Intratumoral Injections of CpG-STAT3 siRNA (CAS3/SS3) in Combination With Local Radiation in Patients With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: CpG-STAT3 siRNA CAS3/SS3 and Localized Radiation Therapy for the Treatment of Relapsed/Refractory B-Cell NHL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: no accrual
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20589; NCI-2021-06965 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20589 (Other: City of Hope Medical Center); P30CA033572 (NIH); P50CA107399 (NIH); Scopus Biopharma (Other: Scopus Biopharma)
Record Dates: First submitted 2021-07-20; First posted 2021-08-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Grade 3b Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Marginal Zone Lymphoma; Refractory Small Lymphocytic Lymphoma; Refractory Grade 3b Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — CPG-oligonucleotide; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (radiation therapy, CAS3/SS3) (Experimental): Patients undergo radiation therapy on days 1 and 2 tumor-bearing lymph node, and receive CAS3/SS3 intratumorally on days 2, 4, 16, and 18. Patients assigned to dose level 3 also receive CAS3/SS3 intratumorally on days 9, 11, 23, and 25.
  Interventions: Biological: CpG-STAT3 siRNA CAS3/SS3; Radiation: Radiation Therapy

INTERVENTIONS:
Biological: CpG-STAT3 siRNA CAS3/SS3 — Given intratumorally
  Other Names: CAS3/SS3; CpG ODN/STAT3 siRNA CAS3/SS3; CpG Oligodeoxynucleotide/STAT3 siRNA CAS3/SS3; CpG/Anti-STAT3 siRNA CAS3/SS3; CpG/STAT3 siRNA CAS3/SS3; TLR9 Agonist/STAT3 siRNA Conjugate CAS3/SS3
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial identifies the best dose and side effects of CpG-STAT3 siRNA CAS3/SS3 (CAS3/SS3) in combination with localized radiation therapy in treating patients with B-cell non-Hodgkin lymphoma that has come back (relapsed) or does not respond to treatment (refractory). CAS3/SS3 simultaneously targets two molecules, TLR9 receptor and STAT3. This investigational drug combines a CpG oligonucleotide and an siRNA in one molecule that act together to interfere with the ability of the cancer cells to grow. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Giving CAS3/SS3 with localized radiation therapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the recommended phase 2 dose (RP2D) of CAS3/SS3 when given in combination with local fixed-dose radiation therapy (RT).

II. Evaluate the safety and feasibility of intratumoral injections of CAS3/SS3 when combined with local fixed-dose RT, by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration.

SECONDARY OBJECTIVES:

I. Characterize the clinical activity (overall and per dose level) of CAS3/SS3 through the assessment of disease response, and response duration. (Clinical) II. Characterize the biologic activity (overall and per dose level) of CAS3/SS3 when combined with local fixed-dose RT by assessing. (Biologic [Immunologic Correlative Studies]) IIa. Silencing of the STAT3 gene and its key downstream genes. IIb. Local and systemic immune responses, including: evidence/extent of immune cell intratumoral infiltration, immune cell activation within the tumor and in the peripheral blood, and changes in proinflammatory mediators in plasma.

OUTLINE:

Patients undergo radiation therapy on days 1 and 2 tumor-bearing lymph node, and receive CAS3/SS3 intratumorally on days 2, 4, 16, and 18. Patients assigned to dose level 3 also receive CAS3/SS3 intratumorally on days 9, 11, 23, and 25.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Age 18 and older
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (corresponds to Karnofsky Performance Status [KPS] of >= 70)
* Life expectancy greater than 16 weeks
* Relapsed/refractory disease; patients must have failed >= 2 prior systemic therapies and have no treatment options known to provide clinical benefit
* Biopsy confirmed relapsed or refractory B-cell lymphoma of the following subtypes; patients with a partial response to a previous treatment are allowed.

  * Follicular grade 1 or 2, or 3 marginal zone or small lymphocytic lymphoma
  * Diffuse large B-cell lymphoma, non-germinal center B-cell like (GCB) type determined by immunohistochemistry using Han's algorithm
  * Mantle cell lymphoma
* Patients must have at least two separate tumor sites, one of which is at least 2 cm in diameter and peripherally accessible and amenable for intratumoral injection of CAS3/SS3 with stabilization by palpation, and the other is at least 1.5 cm in diameter
* Tumor specimens must be available for immunological studies either from a previous biopsy or a new biopsy obtained before the initiation of the study. Paraffin-embedded specimens are acceptable
* Required wash out periods for prior therapy:

  * Topical therapy: 2 weeks
  * Chemotherapy: 4 weeks
  * Radiotherapy: 4 weeks
  * Other investigational therapy: 4 weeks
  * Monoclonal antibody or immunotherapy: 4 weeks
  * Targeted therapies: 4 weeks
  * Allogeneic transplant: 6 months
* Absolute neutrophil count (ANC) >= 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin >= 8 g/dl
* Total serum bilirubin (mg/dL): =< 1.5 x upper normal limit (ULN)
* Aspartate aminotransferase (AST) < 3 x ULN without liver metastasis and < 5 x ULN with liver metastasis
* Alanine aminotransferase (ALT) < 3 x ULN without liver metastasis and < 5 x ULN with liver metastasis
* Adequate renal function as determined by serum creatinine =< 2.0 mg/dL or creatinine clearance of >= 50 mL/min per the Cockcroft-Gault formula
* International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Female of childbearing potential: serum pregnancy test
* Cardiac function 12-lead electrocardiogram (ECG) to confirm the absence of clinically significant arrhythmias
* Left ventricular ejection fraction (LVEF) >= 45%
* Oxygen saturation on room air of >= 92%
* The effects of CAS3/SS3 on the developing fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Patients may not be receiving any other investigational agents, or concurrent biological, chemotherapy, or radiation therapy
* Current use of anticoagulant therapy (aspirin [ASA] =< 325 mg per day allowed) or history of significant bleeding diathesis
* Treatment with corticosteroids or other systemic immunosuppressive medication (e.g., methotrexate, rapamycin) within 28 days of study treatment. Note: patients with adrenal insufficiency may take up to 7.5 mg of prednisone or equivalent daily. Topical and inhaled corticosteroids in standard doses are allowed
* Patients with rapid progression of disease requiring immediate anti lymphoma therapy
* Patients should not have any uncontrolled illness including ongoing or active infection
* Pregnant or lactating women are excluded from this study because CAS3/SS3is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAS3/SS3, breastfeeding should be discontinued if the mother is treated with CAS3/SS3
* Prior malignancy (active within 5 years of screening) except basal cell or completely excised non-invasive squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix
* Pre-existing autoimmune or antibody mediated disease including: systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, Addison's disease, but excluding the presence of autoantibodies without clinical autoimmune disease
* History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, or current acute colitis of any origin
* History of diverticulitis (even a single episode) or evidence of diverticulitis at baseline, including evidence limited to computed tomography (CT) scan only. Note: diverticulosis is not an exclusion criterion per se
* Graft versus host disease
* Severe psoriasis
* Active thyroiditis
* History of uveitis
* Known history of human immunodeficiency virus (HIV) with detectable viral load or patients with acquired immuno-deficiency syndrome (AIDS) are excluded
* Known active or chronic viral hepatitis B or C infection
* Patients with active infection or with a fever > 38.5 degrees Celsius (C) within three days prior to the first scheduled treatment
* Active central nervous system (CNS) metastases
* History of allergic reactions attributed to compounds of similar composition to agatolimod sodium (PF-3512676) or tremelimumab
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to CAS3/SS3
* Significant cardiovascular disease (i.e. New York Heart Association [NYHA] >= class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias)
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 6 months
  Toxicity will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5. Observed toxicities will be summarized in terms of type (organ affected or laboratory determination), severity, attribution, time of onset, duration, and reversibility or outcome.
Dose Limiting Toxicity | Up to 56 days
  Grade 3 or higher toxicities at least possibly related to study treatment as assessed by CTCAE, with noted exceptions.

SECONDARY OUTCOMES:
Overall response | From 56 days through 6 months
  Will be categorized using the 2014 Lugano response criteria for malignant lymphoma.
Response duration | Up to 6 months
  Time interval from the date of first documented response (CR or PR) to documented disease relapse, progression or death whichever occurs first, assessed up to 2 years
Suppression of STAT3 expression | up to 56 days
  Measurement of STAT3 mRNA cleavage in lymph node tissue and peripheral blood mononuclear cells using RACE
Suppression of STAT3 activation of downstream targets. | Up to 19 days
  Suppression of STAT3 activation of downstream target genes and immune genes as assessed by Nanostring in lymph node tissue
Activation of immune cells | Up to 56 days
  Serum IFNs, IP-10, MCP1 levels will be evaluated as evidence for systemic effects of CAS3/SS3 injections.

CONTACTS AND LOCATIONS:
Overall Officials: Lihua E Budde, Principal Investigator — City of Hope Medical Center